CLINICAL TRIAL: NCT02355028
Title: A Randomized, Double-Masked, Vehicle-Controlled Proof-Of-Concept Study for Topically Delivered LHA510 as a Maintenance Therapy in Patients With Wet Age-Related Macular Degeneration (AMD)
Brief Title: LHA510 Proof-of-Concept Study as a Maintenance Therapy for Patients With Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LHA510-2201
Record Dates: First submitted 2015-01-28; First posted 2015-02-04 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-11

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: LHA510; PoC; Age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — acrizanib; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LHA510 (Experimental): LHA510 ophthalmic suspension administered topically in the study eye as specified in the protocol for 84 days, with ranibizumab ophthalmic solution for IVT injection as standard of care rescue therapy.
  Interventions: Drug: LHA510 ophthalmic suspension; Drug: Ranibizumab ophthalmic solution
- Vehicle (Placebo Comparator): LHA510 vehicle administered topically in the study eye as specified in the protocol for 84 days, with ranibizumab ophthalmic solution for IVT injection as standard of care rescue therapy.
  Interventions: Drug: LHA510 vehicle; Drug: Ranibizumab ophthalmic solution

INTERVENTIONS:
Drug: LHA510 ophthalmic suspension
  Arms: LHA510
Drug: LHA510 vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle
Drug: Ranibizumab ophthalmic solution — For intravitreal (IVT) injection
  Other Names: Lucentis®

SUMMARY:
The purpose of this study is to evaluate the efficacy of 84 successive days of topically administered LHA510 compared to vehicle in reducing the number of patients requiring intravitreal (IVT) anti-vascular endothelial growth factor (VEGF) therapy (Lucentis®) for recurrence of active choroidal neovascularization (CNV).

DETAILED DESCRIPTION:
On Day -1, patients will receive an IVT Lucentis® injection in the study eye, and then will be randomized to receive either topical LHA510 ophthalmic suspension or vehicle in a 1:1 ratio for 84 days. Patients with recurrence of active CNV in the study eye during the study will receive rescue IVT Lucentis® injections. Following the treatment period, subjects will return for a follow-up visit and a disposition visit. Only one eye (designated as the study eye) will be dosed with either topical LHA510 or vehicle per patient.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent form;
* Wet AMD;
* IVT anti-VEGF therapy for at least 6 months and a maximum of 7 years since the 3rd loading dose;
* BCVA 50 letters (approximate Snellen equivalent 20/100) or better in the study eye;
* Demonstrate ability to administer eye drops (subject or care-giver);
* CNV recently demonstrated high need for frequent anti-VEGF therapy and a sustained functional and clear anatomical response to the therapy in the study eye;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any active ocular or periocular infection or intraocular inflammation;
* Current or history of macular or retinal disease (if visually significant) other than wet AMD in the study eye;
* Current clinically significant vitreous hemorrhage or history of rhegmatogenous retinal detachment affecting the macula in the study eye;
* History of hypersensitivity to any of the study drugs or clinically relevant sensitivity to fluorescein dye or povidone iodine;
* Women of child-bearing potential;
* History of a medical condition that, in the opinion of the Investigator, would preclude scheduled study visits, completion of the study or a safe administration of investigational product;
* Other protocol-specified exclusion criteria may apply.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Scientist, CA CSI, ID/Multi-TA, Study Director — Novartis Institutes for BioMedical Research, Inc.
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 20 study centers located in the United States.
Pre-assignment Details: Of the 136 enrolled, 37 subjects were exited as screen failures and another 6 subjects were discontinued prior to randomization. This reporting group includes all randomized subjects (93).
Period: Overall Study
Arm/Group | LHA510 | Vehicle
Started | 47 | 46
Treated | 46 | 45
Completed | 36 | 41
Not Completed | 11 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Deemed ineligible after randomization | 8 | 4

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who received any dose of investigational product (IP) (Safety Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | LHA510 | Vehicle | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (7.74) | 76.8 (7.94) | 77.1 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 24 | 17 | 41
Central Subfield Thickness Total (CSFTtot) [Mean (Standard Deviation); unit: μm] — The thickness of the retina was measured using spectral domain-optical coherence tomography (SD-OCT) and reported in micrometers. Population: All subjects who met amendment 4 entry criteria, received any dose of IP, had at least 1 follow-up visit with an assessment for primary endpoint, and had no critical protocol deviations, or discontinued the study due to lack of efficacy or tolerability before Day 84 (Extended PPS-A4).
  μm
    number analyzed (Participants) | 33 | 37 | 70
    (all) | 350.5 (107.09) | 374.9 (116.98) | 363.4 (112.29)
Best-corrected visual acuity (BCVA) [Mean (Standard Deviation); unit: letters] — Measurement of best corrected (with spectacles or other visual corrective devices) visual acuity was conducted in each eye individually using Early Treatment Diabetic Retinopathy Study (ETDRS) charts and reported in number of letters read correctly. Population: Extended PPS-A4
  letters
    number analyzed (Participants) | 33 | 37 | 70
    (all) | 71.2 (9.45) | 70.5 (8.87) | 70.9 (9.09)
Central Subfield Thickness Neuro-Retina (CSFTnr) [Mean (Standard Deviation); unit: μm] — The thickness of the neuro-retina, at the level of the central subfield, was measured using SD-OCT and reported in micrometers. Population: Extended PPS-A4
  μm
    number analyzed (Participants) | 33 | 37 | 70
    (all) | 242.2 (48.95) | 239.0 (75.87) | 240.5 (64.17)
Lesion Thickness [Mean (Standard Deviation); unit: μm] — The thickness of the neovascular lesion was measured using SD-OCT and reported in micrometers. Population: Extended PPS-A4
  μm
    number analyzed (Participants) | 33 | 37 | 70
    (all) | 20.3 (37.90) | 45.8 (92.83) | 33.8 (72.99)
Subretinal Fluid-Foveal Involvement (SRFfi) Thickness [Mean (Standard Deviation); unit: μm] — The thickness of subretinal fluid involving the fovea was measured using SD-OCT and reported in micrometers. Population: Extended PPS-A4
  μm
    number analyzed (Participants) | 33 | 37 | 70
    (all) | 40.7 (58.81) | 25.0 (50.76) | 32.4 (54.87)
Pigment Epithelial Detachment - Foveal Involvement (PEDfi) Thickness [Mean (Standard Deviation); unit: μm] — The thickness of pigment epithelial detachment involving the fovea was measured using SD-OCT and reported in micrometers. Population: Extended PPS-A4
  μm
    number analyzed (Participants) | 33 | 37 | 70
    (all) | 60.9 (92.26) | 82.6 (100.07) | 72.4 (96.39)
Total Lesion Size [Mean (Standard Deviation); unit: mm^2] — The total neovascular lesion size was measured by fluorescein angiography (FA) assessment and reported in millimeters squared. Population: Extended PPS-A4
  mm^2
    number analyzed (Participants) | 32 | 35 | 67
    (all) | 6.1 (4.73) | 7.8 (5.74) | 7.0 (5.31)
Choroidal Neovascularization (CNV) Size [Mean (Standard Deviation); unit: mm^2] — CNV (creation of new blood vessels in the choroid layer of the eye) size as measured by FA assessment and reported in millimeters squared. Population: Extended PPS-A4
  mm^2
    number analyzed (Participants) | 32 | 35 | 67
    (all) | 6.0 (4.79) | 7.7 (5.72) | 6.9 (5.33)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Positive LUCENTIS® Retreatment Status at Day 84
Description: For subjects who completed the Day 84 visit, retreatment need status was positive if LUCENTIS® retreatment (injection) was required before or at Day 84, including requiring retreatment at or before the Day 84 visit with the actual retreatment performed at a later visit.
Time Frame: Day 84
Population: Extended PPS-A4
Measure: Count of Participants; unit: Participants
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
Participants | 25 | 25

2. Secondary Outcome: Time to First LUCENTIS® Retreatment Need Identification up to Day 84
Description: The time was determined based on the visit of the treatment period when a patient was identified as requiring retreatment with LUCENTIS.
Time Frame: Day 14, Day 28, Day 56, Day 84
Population: Extended PPS-A4 who required retreatment
Measure: Count of Participants; unit: Participants
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 25 | 25
Participants
  Day 14 | 0 | 0
  Day 28 | 5 | 8
  Day 56 | 16 | 11
  Day 84 | 4 | 6

3. Secondary Outcome: Number of LUCENTIS® Retreatment Needs Identified Required up to Day 84
Description: The number of LUCENTIS retreatment needs identified before or at the Day 84 visit (even if retreatment was applied at a later visit) for each patient was used in the analysis
Time Frame: Up to Day 84
Population: Extended PPS-A4
Measure: Number; unit: participants
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
participants
  0 retreatment injections | 8 | 12
  1 retreatment injection | 18 | 18
  2 retreatment injections | 6 | 6
  3 retreatment injections | 1 | 1

4. Secondary Outcome: Number of Subjects Requiring LUCENTIS® Retreatment at Days 28 and 56
Description: The number of LUCENTIS® retreatment needs identified before or at the Day 28 and Day 56 visits (even if retreatment was applied at a later visit) for each subject was used in the analysis.
Time Frame: Day 28, Day 56
Population: Extended PPS-A4
Measure: Count of Participants; unit: Participants
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
Participants
  Day 28 | 5 | 8
  Day 56 | 21 | 19

5. Secondary Outcome: Change From Randomization Visit (Day -1) in Central Subfield Thickness Total (CSFTtot) at All Visits at the Study Site
Description: The thickness of the retina was measured using SD-OCT and reported as a difference, in micrometers, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction in thickness, whereas a positive number indicates an increase. An increase in thickness may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 14, Day 28, Day 56, Day 84
Population: Extended PPS-A4. Missing data imputed using the Last Observation Carried Forward (LOCF) approach.
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
μm
  Day 14 | -46.9 (8.40) | -43.0 (7.93)
  Day 28 | -38.6 (7.42) | -28.9 (7.00)
  Day 56 | 11.3 (10.01) | 1.0 (9.45)
  Day 84 | -16.8 (8.92) | -12.2 (8.42)

6. Secondary Outcome: Change From Randomization Visit (Day -1) in Best Corrected Visual Acuity (BCVA) at All Visits at the Study Site
Description: Measurement of best corrected (with spectacles or other visual corrective devices) visual acuity was conducted in each eye individually using ETDRS charts and reported in number of letters read correctly. An increase (gain) in letters read from the baseline assessment indicates improvement. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 14, Day 28, Day 56, Day 84
Population: Extended PPS-A4. Missing Data Imputed Using LOCF.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
letters
  Day 14 | 1.3 (0.80) | 1.6 (0.75)
  Day 28 | 1.7 (0.89) | 2.5 (0.84)
  Day 56 | -0.5 (1.28) | 2.3 (1.21)
  Day 84 | -1.7 (1.59) | 2.2 (1.50)

7. Secondary Outcome: Change From Randomization Visit (Day -1) in Central Subfield Thickness, Neuro-retina (CSFTnr) by Visit
Description: The thickness of the neuro-retina, at the level of the central subfield, was measured using SD-OCT and reported as a difference, in micrometers, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction in thickness, whereas a positive number indicates an increase. An increase in thickness may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 28, Day 84
Population: Extended PPS-A4. Missing data imputed using LOCF.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
μm
  Day 28 | -16.6 (22.62) | -15.1 (38.21)
  Day 84 | -4.1 (35.34) | -8.8 (36.75)

8. Secondary Outcome: Change From Randomization Visit (Day -1) in Lesion Thickness by Visit
Description: The thickness of the neovascular lesion was measured using SD-OCT and reported as a difference, in micrometers, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction in thickness, whereas a positive number indicates an increase. An increase in thickness of the neovascular lesion may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 28, Day 84
Population: Extended PPS-A4. Missing data imputed using LOCF.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
μm
  Day 28 | -1.9 (38.05) | 6.9 (43.66)
  Day 84 | 1.4 (26.46) | 6.9 (43.96)

9. Secondary Outcome: Change From Randomization Visit (Day -1) in Subretinal Fluid - Foveal Involvement (SRFfi) Thickness by Visit
Description: The thickness of subretinal fluid involving the fovea was measured using SD-OCT and reported as a difference, in micrometers, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction in thickness, whereas a positive number indicates an increase. An increase in thickness of subretinal fluid involving the fovea may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 28, Day 84
Population: Extended PPS-A4. Missing Data Imputed Using LOCF.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
μm
  Day 28 | -18.5 (44.67) | -11.0 (34.73)
  Day 84 | -14.1 (54.08) | -5.9 (31.33)

10. Secondary Outcome: Change From Randomization Visit (Day -1) in Pigment Epithelial Detachment - Foveal Involvement (PEDfi) Thickness by Visit
Description: The thickness of pigment epithelial detachment involving the fovea was measured using SD-OCT and reported as a difference, in micrometers, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction in thickness, whereas a positive number indicates an increase. An increase in thickness of pigment epithelial detachment involving the fovea may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 28, Day 84
Population: Extended PPS-A4. Missing Data Imputed Using LOCF.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 33 | 37
μm
  Day 28 | -0.3 (38.92) | -13.3 (43.23)
  Day 84 | -0.2 (33.33) | -7.6 (47.25)

11. Secondary Outcome: Change From Randomization Visit (Day -1) in Total Lesion Size by Visit
Description: The total wet AMD lesion size was measured using FA and reported as a difference, in millimeter squared, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction, whereas a positive number indicates an increase. An increase in wet AMD lesion size may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 84
Population: Extended PPS-A4 as observed
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 32 | 35
mm^2 | -0.3 (1.71) | 0.5 (1.81)

12. Secondary Outcome: Change From Randomization Visit (Day -1) in CNV Size by Visit
Description: The size of CNV (area of new blood vessels in the choroid layer of the retina) was measured using FA and reported as a difference, in millimeter squared, between a given post-Randomization Visit and Randomization Visit (Day-1). A negative number indicates a reduction, whereas a positive number indicates an increase. An increase in CNV size may indicate a progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Day -1, Day 84
Population: Extended PPS-A4 as observed
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | LHA510 | Vehicle
Number analyzed (Participants) | 32 | 35
mm^2 | -0.6 (2.00) | 0.5 (1.71)

13. Secondary Outcome: Plasma Concentration of LHA510 and CRA398
Description: Samples collected from subjects, after multiple topical ocular dosing of LHA510, were analyzed to determine concentrations of LHA510 and its metabolite, CRA398. Plasma LHA510 and CRA398 concentrations were quantitated by a validated liquid chromatography-tandem mass spectroscopy assay method. Below the limit of quantification (BLQ) is treated as zero.
Time Frame: Day 28, Day 84
Population: This analysis population includes all subjects who were treated with LHA510, had at least 1 serum sample following exposure to the IP, and had no known specimen collection or analytical deviations, as identified by the Pharmacokineticist, that would have affected the integrity of the data [Pharmacokinetics (PK) Analysis Set].
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- LHA510: LHA510 dose twice daily (BID) by Day 28, LHA510 dose once daily (QD) by Day 84, LHA510 dose 3-times daily (TID) by Day 84
- CRA398: Metabolite of LHA510
Arm/Group | LHA510 | CRA398
Number analyzed (Participants) | 31 | 31
ng/mL
  Day 28, BID | 0.0746 (0.0483) | 0.0257 (0.0287)
  Day 84, QD: number analyzed (Participants) | 6 | 6
  Day 84, QD | 0.0403 (0.0225) | 0 (0)
  Day 84, TID: number analyzed (Participants) | 10 | 10
  Day 84, TID | 0.0694 (0.0439) | 0.0160 (0.0179)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 177 days). AEs are reported as pre-treatment, treatment-emergent, and post-treatment.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered a study treatment regardless of whether or not the event had a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: All subjects with AE/s reported prior to the initiation of IP administration
- LHA510; Vehicle: All subjects with AE/s having an onset from IP initiation and up through 7 days after cessation of IP administration
- Post-treatment LHA510; Post-treatment Vehicle: All subjects with AE/s having an onset more than 7 days after IP administration cessation through the study exit
Arm/Group | Pre-treatment | LHA510 | Vehicle | Post-treatment LHA510 | Post-treatment Vehicle
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/46 | 0/45 | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/136 | 1/46 | 0/45 | 1/46 | 0/45
Other Adverse Events (participants affected / at risk) | 1/136 | 28/46 | 5/45 | 3/46 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=136) | LHA510 (N=46) | Vehicle (N=45) | Post-treatment LHA510 (N=46) | Post-treatment Vehicle (N=45)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=136) | LHA510 (N=46) | Vehicle (N=45) | Post-treatment LHA510 (N=46) | Post-treatment Vehicle (N=45)
Corneal oedema (Eye disorders) | 0 | 8 | 0 | 0 | 0
Corneal opacity (Eye disorders) | 0 | 20 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 5 | 3 | 0 | 0
Eye pain (Eye disorders) | 1 | 3 | 0 | 0 | 0
Keratopathy (Eye disorders) | 0 | 5 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 6 | 1 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 3 | 0 | 0 | 0
Vital dye staining cornea present (Investigations) | 0 | 4 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.